CLINICAL TRIAL: NCT03740568
Title: Effect of Intervention on Progesterone Levels Before Euploid Embryo Transfer in Pregnancy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Collaborators: Fundación Santiago Dexeus Font (Other); Dexeus Clinic Woman (Other)
Responsible Party: Principal Investigator, Buenaventura Coroleu, Head Reproductive Service, Fundacion Dexeus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-PRG-2018-09
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Infertility; Progesterone; Frozen Embryo Transfer; Euploid Embryo Transfer; Pregnancy Outcome; Artificial Cycle; Ongoing Pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Progesterone group (Other): Progesterone level >10.64 ng/mL on day 4 of progesterone supplementation
  Interventions: Drug: Normal Progesterone
- Low Progesterone group (Experimental): Progesterone level <10.64 ng/mL on day 4 of progesterone supplementation
  Interventions: Drug: Low Progesterone

INTERVENTIONS:
Drug: Low Progesterone — Additional daily dosage of subcutaneous progesterone (Psc) 25 mg/day at night since D4 (vaginal micronized P 200mg/200mg/200mg + Psc 25 mg/night) New Progesterone analysis on D5 before warming the embryo. Group 2a (Canceled Group, P on D5 <10.64 ng/mL): cancel PGT-FET. Scheduling a new procedure under different P supplementation.
  Group 2b (Restored Progesterone Group, P on D5 >10.64 ng/mL): continue HRT as previously described (vaginal micronized P 200mg/200mg/200mg + Psc 25 mg/night). Warming and transfer the same day (D5)
  Beta-hCG and P analysis is performed on the 14th day of P supplementation (D14). In case of positive Beta-hCG analysis:
  If P is >10.64 ng /mL: the same P supplementation is continued. If P is <10.64 ng /mL: an additional dosage of vaginal micronized P (200 mg) is added at night
  Arms: Low Progesterone group
Drug: Normal Progesterone — Same Progesterone supplementation (vaginal micronized P 200mg/200mg/200mg) Warming and transfer on D5
  Beta-hCG and P analysis is performed on the 14th day of P supplementation (D14). In case of positive Beta-hCG analysis:
  If P is >10.64 ng /mL: the same P supplementation is continued. If P is <10.64 ng /mL: an additional dosage of vaginal micronized P (200 mg) is added at night
  Arms: Normal Progesterone group

SUMMARY:
Transferring an euploid embryo avoids one of the main reasons of miscarriage and implantation failure (1), overcoming confounding factors such as embryo ploidy or maternal age. Frozen Euploid Embryo Transfer (FEET) is routinely performed under standard hormone replacement therapy (HRT) and could be considered the best model for evaluating the impact of the endometrial preparation in clinical pregnancy rate and also in miscarriage rate.

Recently several authors have paid attention to serum progesterone (P) as a possible factor influencing Frozen Embryo Transfer (FET) outcomes. P plays an important role in endometrial gland formation, embryonic implantation and pregnancy maintenance. Labarta et al. (2) described in blastocyst FET performed under HRT that serum P <9.2 ng/mL measured on the transfer day is associated to significantly lower ongoing pregnancy rate (OR 0.297, 95% CI:0.113-0.779).

Recently the investigators have analyzed 244 FEET performed under HRT in a retrospective study (3). Preimplantation genetic testing for aneuploidies (PGT-A) was carried out as previously described (4). Embryos that reached the blastocyst stage were biopsied and frozen immediately afterwards using the vitrification method (5). Euploid embryos were transferred in a subsequent cycle under HRT. Serum P was analyzed the day previous to FEET. Patients with serum P <10.6 ng/mL had significantly higher miscarriage rate (26.6% vs 9.5%, p=0.007) and lower live birth rate (47.5% vs 62.3 %, p= 0.029) than those with serum P >10.6 ng/mL. The investigators also observed that patients with serum P >13.1 ng/mL had the lowest miscarriage rate (9.1%) and the highest live birth rate (65.6%). The worst outcomes were observed when serum P was <8.06 ng /mL (41% live birth rate and 32.4% miscarriage rate).

As miscarriage was higher among FEET cycles with serum P <10.6 ng/ml, the investigators hypothesize that altering the progesterone supplementation scheme could potentially reduce miscarriage rates and increase live birth rate. The purpose of this study is to modify the standard progesterone supplementation in FEET under HRT (vaginal micronized progesterone 200 mg every 8 hours) (6) according to serum P measured not only on the day prior to transfer but also on Beta subunit of Human Chorionic Gonadotropin (β-hCG) analysis day, and to probe if this intervention reduces miscarriage rate and increases pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* FEET of at least one single embryo
* HRT
* Endometrial thickness >= 6 mm measured day 4 of progesterone supplementation

Exclusion Criteria:

* Patients with mosaic embryos.
* Uterine abnormality.
* Natural cycle protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 598 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Ongoing Pregnancy Rate (OPR) | 12 weeks after transfer procedure
  Ongoing Pregnancy Rate (OPR) beyond pregnancy week 12 in FEET according to serum P level and interventions on D4 and D5
Miscarriage Rate (MR) | 12 weeks after transfer procedure
  Miscarriage Rate (MR) in FEET according to serum P level and interventions on D4 and D5.
Concentration of serum P level | D4, D5 and D14 of P supplementation
  P level

SECONDARY OUTCOMES:
Rate of cancellation due to lack of response in case of additional Psc dose on D4. | Day 5 of progesterone supplementation
Rate of rescued cycles in case of additional Psc dose | Day 5 of progesterone supplementation
Ongoing Pregnancy Rate and Live Birth Rate according to serum P level and interventions n D14 | On day 14 of progesterone supplementation
Live birth Rate (LBR) | 40 weeks after transfer procedure
  Live birth Rate (LBR) in FEET according to serum P level and interventions on D4 and D5 and D14.

CONTACTS AND LOCATIONS:
Overall Officials: Bueaventura Coroleu, PhD, Study Chair — Hospital Universitari Dexeus. Departamento de Ginecología, Obstetricia y Reproducción
Locations (1):
- Departamento Ginecología, Obstetricia y Reproducción . Hospital Universitari Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubio C, Bellver J, Rodrigo L, Castillon G, Guillen A, Vidal C, Giles J, Ferrando M, Cabanillas S, Remohi J, Pellicer A, Simon C. In vitro fertilization with preimplantation genetic diagnosis for aneuploidies in advanced maternal age: a randomized, controlled study. Fertil Steril. 2017 May;107(5):1122-1129. doi: 10.1016/j.fertnstert.2017.03.011. Epub 2017 Apr 19. PMID 28433371
- [Background] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Corrigendum: Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2018 Jan 1;33(1):178. doi: 10.1093/humrep/dex353. No abstract available. PMID 29177428
- [Background] Gaggiotti-Marre S, Martinez F, Coll L, Garcia S, Alvarez M, Parriego M, Barri PN, Polyzos N, Coroleu B. Low serum progesterone the day prior to frozen embryo transfer of euploid embryos is associated with significant reduction in live birth rates. Gynecol Endocrinol. 2019 May;35(5):439-442. doi: 10.1080/09513590.2018.1534952. Epub 2018 Dec 26. PMID 30585507
- [Background] Coll L, Parriego M, Boada M, Devesa M, Arroyo G, Rodriguez I, Coroleu B, Vidal F, Veiga A. Transition from blastomere to trophectoderm biopsy: comparing two preimplantation genetic testing for aneuploidies strategies. Zygote. 2018 Jun;26(3):191-198. doi: 10.1017/S0967199418000084. Epub 2018 May 25. PMID 29798732
- [Background] Sole M, Santalo J, Boada M, Clua E, Rodriguez I, Martinez F, Coroleu B, Barri PN, Veiga A. How does vitrification affect oocyte viability in oocyte donation cycles? A prospective study to compare outcomes achieved with fresh versus vitrified sibling oocytes. Hum Reprod. 2013 Aug;28(8):2087-92. doi: 10.1093/humrep/det242. Epub 2013 Jun 5. PMID 23744895
- [Background] Martinez F, Boada M, Coroleu B, Clua E, Parera N, Rodriguez I, Barri PN. A prospective trial comparing oocyte donor ovarian response and recipient pregnancy rates between suppression with gonadotrophin-releasing hormone agonist (GnRHa) alone and dual suppression with a contraceptive vaginal ring and GnRH. Hum Reprod. 2006 Aug;21(8):2121-5. doi: 10.1093/humrep/del121. Epub 2006 Apr 21. PMID 16632462
- [Derived] Alvarez M, Gaggiotti-Marre S, Martinez F, Coll L, Garcia S, Gonzalez-Foruria I, Rodriguez I, Parriego M, Polyzos NP, Coroleu B. Individualised luteal phase support in artificially prepared frozen embryo transfer cycles based on serum progesterone levels: a prospective cohort study. Hum Reprod. 2021 May 17;36(6):1552-1560. doi: 10.1093/humrep/deab031. PMID 33686413
- See also: Related Info — https://www.dexeus.com/